CLINICAL TRIAL: NCT05851898
Title: The Role of SNRI's in the Prophylaxis of Depression in the First Year Following Lower Extremity Fragility Fractures in Geriatric Patients
Brief Title: Serotonin-norepinephrine Reuptake Inhibitor in Prophylaxis of Depression Following Fragility Fractures
Acronym: SNRI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00095504
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Depression in Old Age; Fragility Fracture
Keywords: Geriatrics; Serotonin-norepinephrine
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: geriatric patients with operative lower extremity fragility fractures that will be started on Serotonin-norepinephrine reuptake inhibitor (SNRI) medication immediately after obtaining consent at index hospitalization or first post operative clinic appointment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Duloxetine 30mg (Experimental): Duloxetine 30mg daily 90 day supply and 3 refills
  Interventions: Drug: Duloxetine 30 mg

INTERVENTIONS:
Drug: Duloxetine 30 mg — Duloxetine 30mg daily prescribed at discharge
  Other Names: Common brands: Irenka, Cymbalta

SUMMARY:
The goal of this pilot study is to learn about the feasibility about prescribing anti-depressants at discharge in patients aged 50 years and older with a lower extremity fragility fracture. The main questions it aims to answer are:

* What are the obstacles to enrolling patients and prescribing anti-depressants among older adults?
* Is it possible to start prescribing SNRI medication upon discharge?
* What is the prevalence of depressive symptoms amongst patients with different types of injuries and weightbearing status?
* What is a transition of care plan for patients who have geriatric depression and require further care?

Participants will:

* Undergo screening using the Geriatric Depression Scale
* Start on Duloxetine 30mg daily at time of discharge
* Report medication compliance and complete re-screening monthly
* Complete patient reported outcome measures and 3 months, 6 months, and 1 year
* Receive a referral to behavioral health, primary care, or psychiatrist for evaluation if they screen positive at any timepoint

DETAILED DESCRIPTION:
As with many mental health diagnoses, there continues to be a stigma against receiving treatment and potentially even more so receiving prophylaxis16. Identifying these hurdles at the patient level will allow us to better educate patients and physicians about the benefits of this intervention. Secondly, this pilot study will help us determine if it is possible to start prescribing SNRI medication upon discharge. It will allow us to navigate the procurement of medications through Medicare, prescribing practices at discharge and address patient concerns regarding starting a new medication.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric (greater than or equal to 65 years old)
* Lower extremity fragility fractures managed operatively

Exclusion Criteria:

* Polytrauma
* Pathological fractures
* Patients on hospice
* Patients with previously diagnosed psychiatric disorders
* Patients with previously diagnosed dementia
* Patients already taking Selective serotonin reuptake inhibitors (SSRI)s and Serotonin- norepinephrine reuptake inhibitors (SNRI)s
* Patients already taking mood stabilizing medication
* Unable to provide informed consent (no use of a legal authorized representative)
* Patients with pre-existing life limiting diagnoses (cancer, etc.)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Geriatric Depression Scale (Short Form) Scores | Baseline
  This scale will be used as the primary outcome in this study as an indicator of patients who develop depression post-operatively. Scores range from 1-15. A score of 5 or greater indicates depression.
Geriatric Depression Scale (Short Form) Scores | up to 1 year
  This scale will be used as the primary outcome in this study as an indicator of patients who develop depression post-operatively. Scores range from 1-15. A score of 5 or greater indicates depression.

SECONDARY OUTCOMES:
PROMIS-29 Subscale Scores - Depression | Month 3, Month 6, and Year 1
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means higher depression.
PROMIS-29 Subscale Scores - Physical Function | Month 3, Month 6, and Year 1
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Possible scores range from 0 to 100, with higher scores representing better health status
Number of patients who have side effects from the medication | Baseline, monthly up to 1 year
  Number of patients who have side effects from the medication
Number of participants who undergo re-operation | Baseline, monthly up to 1 year
  Number of participants who undergo re-operation
Number of participants who are readmitted to the hospital | Baseline, monthly up to 1 year
  Number of participants who are readmitted to the hospital
Mortality Rate | Baseline, monthly up to 1 year
  Mortality Rate
Number of participants who re-fracture the study injury | Baseline, monthly up to 1 year
  Number of participants who re-fracture

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Seymour, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No